CLINICAL TRIAL: NCT03537742
Title: PCSK9 Inhibition After Heart Transplantation
Brief Title: Cardiac Allograft Vasculopathy Inhibition with Alirocumab
Acronym: CAVIAR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, William Fearon, Professor, Cardiovascular Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-45975; 4R33HL139929 (NIH)
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Vasculopathy
Keywords: Heart Transplant
MeSH Terms: conditions — Vascular Diseases | interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- alirocumab (Experimental): alirocumab 150mg subcutaneous every other week for one year following start of study drug
  Interventions: Biological: alirocumab
- placebo (Placebo Comparator): placebo to match alirocumab every other week for one year following start of study drug
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: alirocumab — alirocumab 150mg Subcutaneous
  Other Names: Praluent
  Arms: alirocumab
Biological: placebo — placebo to match alirocumab
  Arms: placebo

SUMMARY:
The focus of this study is to test the safety and efficacy of the PCSK9 inhibitor, alirocumab when administered early after heart transplantation (HT).The main objective of this project is to test the safety and impact on cardiac allograft vasculopathy (CAV) of alirocumab when given early after HT.

ELIGIBILITY:
Inclusion Criteria:

* Heart Transplant recipient

Exclusion Criteria:

* impaired liver function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-05-13 (Actual); Primary Completion 2025-07-28 (Estimated); Study Completion 2025-08-28 (Estimated)

PRIMARY OUTCOMES:
Change in volume of plaque at 1 year post study drug start post heart transplant | Baseline and one year
  Measured change in coronary artery plaque volume(MM3), measured by Intravascular Ultrasound at time of coronary arteriogram within 4-8 weeks post transplant( baseline) and one year after study drug start post transplant

SECONDARY OUTCOMES:
Change in LDL-C | Baseline, 3, 6 and 12 months
  measure differences in LDL-C lipid particle values between the two arms at baseline, 3, 6 and 12 months
Change in lipoprotein (a) | Baseline, 3, 6 and 12
  measure differences lipid particle lipoprotein (a) values between the two arms at Baseline, 3, 6 and 12 months
Change in apolipoprotein B | Baseline, 3, 6 and 12
  measure differences in apolipoprotein B lipid particle apolipoprotein B values between the two arms at baseline, 3, 6 and 12 months
Percent change in coronary vessel size by fractional flow reserve | baseline and one year
  evaluate the ability of fractional flow reserve (% change in vessel size) to predict clinically meaningful increases in plaque volume one year post-transplant relative to that of plaque volume measured via intravascular ultrasound at baseline

CONTACTS AND LOCATIONS:
Overall Officials: William F Fearon, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fearon WF, Terada K, Takahashi K, Skoda A, Luikart HI, Lamendola CA, Zimmermann FM, Hashikata T, Saito K, Yoshida A, Varr B, Knowles JW, Woo C, Honda Y, Teuteberg J, Khush KK. Cardiac Allograft Vasculopathy Inhibition With Alirocumab: The CAVIAR Trial. Circulation. 2026 Jan 6;153(1):7-17. doi: 10.1161/CIRCULATIONAHA.125.077603. Epub 2025 Nov 10. PMID 41212178